CLINICAL TRIAL: NCT03592732
Title: The Impact Of Adipokines Levels In Patients With Atrial Fibrillation
Brief Title: The Role of Adipokines In Atrial Fibrillation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Maria Velliou, Principal Investigator, University of Athens
Other Study IDs: 308/29-3-2018
Record Dates: First submitted 2018-06-28; First posted 2018-07-19 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Atrial Fibrillation; Adiposity; Adiponectin; Visceral Obesity; Hormone Disturbance
MeSH Terms: conditions — Atrial Fibrillation; Obesity; Obesity, Abdominal; Endocrine System Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A: Patients with atrial fibrillation
  Interventions: Other: Blood sample
- B: Patients without atrial fibrillation
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Blood sample

SUMMARY:
The principal aim of the present study is to analyze adiponectin, omentin-1, apelin and visfatin plasma levels in patients with and without AF in an effort to identify their potential role in the development of AF.

DETAILED DESCRIPTION:
Introduction Adipose tissue is no longer considered a triglycerides-storage depot, but it has been recognized as an endocrine organ that regulates sugar and fat metabolism and energy homeostasis and implicates in cardiovascular (CV) function through the release of bioactive factors, the so-called adipokines. Several adipokines including adiponectin, omentin-1, apelin and visfatin have been identified as well as their link with CV diseases and, particularly, coronary artery disease (CAD) (1-3).

However, the potential impact of adipokines in patients with atrial fibrillation (AF) has not still elucidated. Although, there is evidence that apelin (4,5) and omentin-1 (6) are inversely correlated with AF, available data in regard to adiponectin and visfatin are inconclusive (7-9).

Objectives The principal aim of the present study is to calculate adiponectin, omentin-1, apelin and visfatin plasma levels in patients with AF and controls matched for age and gender in an effort to identify their potential role in the development of AF.

Methods Study population. Overall, 40 patients with AF and 40 controls will be studied. Patients with CAD, heart failure, cardiomyopathy, cancer, significant valvular disease, rheumatic heart disease or stroke will be excluded. The present study is conducted in accordance with the Declaration of Helsinki and has been approved by the Ethics Committee of our Hospital. A written informed consent will be obtained from each participant.

A detailed profile including demographic characteristics (age, gender) and traditional CV risk factors (smoking, hypertension, dyslipidemia, diabetes mellitus) will be obtained from every patient. Body mass index was (BMI) will be calculated as bodyweight in kilograms divided by height in meters squared and will be estimated for all subjects. All participants will undergo either electrocardiogram or 24-hour Holter monitoring. AF patients will be divided into the following three groups: paroxysmal AF, persistent AF and permanent AF.

Definitions. Paroxysmal AF is defined as a history of one or more episodes of AF that were treated with pharmacological or electrical cardioversion within seven days. Persistent AF is defined a history of one or more episodes of AF over seven days that required pharmacological or electrical cardioversion) and permanent AF is defined as continuous AF for more than a year.

Echocardiography. Transthoracic echocardiography will be performed in every patient. Left atrial dimension, interventricular septal dimension, left ventricular (LV) end diastolic dimension and ejection fraction (EF) will be measured.

Laboratory analysis. Blood samples will be collected after 12-hour overnight fasting. Plasma adiponectin (RD195023100,Human Adiponectin, Elisa Bio Vendor Laboratory, Medicine Inc., Brno, Czech Republic), omentin-1, apelin (Phoenix Pharmaceuticals Inc, Burlingame, CA) and visfatin (Phoenix Pharmaceuticals, California, CA, USA) levels will be measured by the Elisa method. Natriuretic peptide, C-reactive protein (CRP) and parameters concerning lipid profile (total cholesterol, triglycerides, low-density cholesterol, high-density cholesterol), glycemic profile (plasma glucose, hemoglobin A1c) and renal function (urea, creatinine) will be measured by standardized enzymatic methods as well.

Statistical analysis. Continuous variables will be expressed as mean values ± standard deviation (SD). Comparisons of continuous variables will be performed by one-way analysis of variance (ANOVA). Categorical data will be expressed as absolute and relative frequencies. All data will be analyzed using Statistical Package for the Social Sciences (SPSS) version 18.0 and all tests will be 2-tailed with the 5% indicating level of significance.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects without atrial fibrillation and subjects with paroxysmal, persistent or permanent atrial fibrillation

Exclusion Criteria:

* Patients with coronary artery disease, acute coronary syndrome, heart failure (EF<50%), cardiomyopathy, cancer, significant valvular disease, rheumatic heart disease, chronic kidney disease (eGRF<30) or stroke will be excluded.

Max Age: 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All participants will undergo either electrocardiogram or 24-hour Holter monitoring. AF patients will be divided into the following three groups: paroxysmal AF, persistent AF and permanent AF.Blood samples will be collected after 12-hour overnight fasting. Plasma adiponectin, omentin-1, apelin and visfatin levels will be measured by the Elisa method. Natriuretic peptide, C-reactive protein (CRP) and parameters concerning lipid profile (total cholesterol, triglycerides, low-density cholesterol, high-density cholesterol), glycemic profile (plasma glucose, hemoglobin A1c) and renal function (urea, creatinine) will be measured by standardized enzymatic methods as well. Transthoracic echocardiography will be performed in every patient.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-03-29 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2021-01-29 (Estimated)

PRIMARY OUTCOMES:
adiponectin, omentin-1, apelin and visfatin plasma levels | blood sample collection analysis (day zero
  adiponectin, omentin-1, apelin and visfatin plasma levels calculation by the Eliza method

CONTACTS AND LOCATIONS:
Overall Officials: Elias Sanidas, MD, PhD, Principal Investigator — Dept. of Cardiology, ESH Excellence Center, LAIKO General Hospital, Athens, Greece
Locations (1):
- LAIKO General Hospital, Athens, Greece, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided